CLINICAL TRIAL: NCT06310200
Title: Involvement of the Sphenopalatine Ganglion in Cold Induced Headaches
Brief Title: Sphenopalatine Ganglion Block and Cold Induced Headaches
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Wright State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRB-2023-398
Record Dates: First submitted 2023-10-12; First posted 2024-03-15 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Cold Induced Headache; Brain Freeze; Cold Induced Cephalgia; Headache
MeSH Terms: conditions — Headache | interventions — Lidocaine; Solutions; denatonium; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All besides PI
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intervention Arm (Experimental): Subjects will receive 1 mL of 4% lidocaine (0.5mL in each nostril) administered by intranasal atomization or 0.9% normal saline administered by intranasal atomization.
  Interventions: Drug: Lidocaine Topical 4% Topical Solution
- Placebo Arm (Placebo Comparator): Subjects will receive normal saline placebo mixed with an edible bittering agent added to blind the participant from recognizing the taste of the lidocaine containing solution.
  Interventions: Drug: Bitrex; Drug: normal saline

INTERVENTIONS:
Drug: Lidocaine Topical 4% Topical Solution — Intranasal administration
  Arms: Intervention Arm
Drug: Bitrex — Bittering agent
  Arms: Placebo Arm
Drug: normal saline — Placebo
  Arms: Placebo Arm

SUMMARY:
The primary objective of this study is to determine if a sphenopalatine ganglion (SPG) block, performed through intranasal atomization of 4% lidocaine, is able to prevent cold induced cephalgia ("Brain Freeze"). Secondary objectives will be to determine the degree of decreased pain/duration of brain freeze after sphenopalatine ganglion block

DETAILED DESCRIPTION:
This study will be performed in two phases. The first phase will include a pre-medicated phase where the subjects will be required to rapidly drink up to ½ of a 32 fluid oz icecold slushy to induce a brain freeze. The flavor will be chosen by the participants. The time to onset, intensity, location, and duration of the headache will be recorded. The second phase will commence when the subjects have returned to their normal pain free state, a minimum of 10 minutes has passed since the resolution of the first cold headache, and they feel ready to move to the next phase. The time from complete resolution of the brain freeze to the start of the second phase will be recorded. Any subject that wishes to drop out from the study at this time is free to do so. They may keep their drink and finish it at a more leisurely pace should they choose.

Then the subjects will receive either 1 mL of 4% lidocaine (0.5mL in each nostril) administered by intranasal atomization or 0.9% normal saline administered by intranasal atomization. The normal saline placebo will be mixed with an edible bittering agent added to blind the participant from recognizing the taste of the lidocaine containing solution.

Only participants that experienced a brain freeze in the first phase will be able to move onto the second phase. Each participant will then rapidly drink up to ½ of a 32 fluid oz ice-cold slushy to induce a brain freeze. The time to onset, intensity, location, and duration of the headache will be recorded.

All pain scores will be recorded using a visual analog scale from 0-100 where 0 is no pain and 100 is the worst pain imaginable. We will also record any side effects that the subjects may experience during or shortly after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Wright State University Emergency Medicine (EM) resident physicians and Wright State Boonshoft School of Medicine medical students
* Over the age of 18 years
* Has gotten at least one brain freeze in their life

Exclusion Criteria:

* Individuals who have never gotten a brain freeze
* Anyone who has had any sort of prior trauma to their oro- or nasopharynx or surgery on their oro- or nasopharynx, not to include dental surgery.
* Pregnant patients
* History of allergy to local anesthetic

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Does sphenopalatine ganglion (SPG) block prevent cold induced cephalgia | 5 months
  The primary objective of this study is to determine if a sphenopalatine ganglion block, performed through intranasal atomization of 4% lidocaine, is able to prevent brain freeze. This study will be performed in two phases. The first phase will include a pre-medicated phase where the subjects will be required to rapidly drink up to ½ of a 32 fluid oz icecold slushy to induce a brain freeze. The second phase will commence when the subjects have returned to their normal pain free state, a minimum of 10 minutes has passed since the resolution of the first cold headache. The time from complete resolution of the brain freeze to the start of the second phase will be recorded. Each participant will then rapidly drink up to ½ of a 32 fluid oz ice-cold slushy to induce a brain freeze. The presence or absence of a cold-induced headache will be recorded for each phase.

SECONDARY OUTCOMES:
Degree of pain | 5 months
  Determine the degree of decreased pain after SPG block. All pain scores will be recorded using a visual analog scale from 0-100 where 0 is no pain and 100 is the worst pain imaginable.
Duration of brain freeze | 5 months
  Determine duration of brain freeze after SPG block; measured in minutes and seconds.
Time to onset of headache | 5 months
  Determined in minutes and seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Brian P Murray, DO, Principal Investigator — Wright State University
Locations (1):
- Wright state emergency medicine offices, Dayton, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee JM, Shin TJ. Use of local anesthetics for dental treatment during pregnancy; safety for parturient. J Dent Anesth Pain Med. 2017 Jun;17(2):81-90. doi: 10.17245/jdapm.2017.17.2.81. Epub 2017 Jun 29. PMID 28879335
- [Background] Hensel O, Burow P, Mages S, Wienke A, Kraya T, Zierz S. Increased Blood Flow Velocity in Middle Cerebral Artery and Headache Upon Ingestion of Ice Water. Front Neurol. 2019 Jun 28;10:677. doi: 10.3389/fneur.2019.00677. eCollection 2019. PMID 31316454
- [Background] Binfalah M, Alghawi E, Shosha E, Alhilly A, Bakhiet M. Sphenopalatine Ganglion Block for the Treatment of Acute Migraine Headache. Pain Res Treat. 2018 May 7;2018:2516953. doi: 10.1155/2018/2516953. eCollection 2018. PMID 29862074
- [Background] Bird N, MacGregor EA, Wilkinson MI. Ice cream headache--site, duration, and relationship to migraine. Headache. 1992 Jan;32(1):35-8. doi: 10.1111/j.1526-4610.1992.hed3201035.x. PMID 1555929
- [Background] Morgan A, Romanello G. Use of the Sphenopalatine Ganglion Block to Treat Migraine Headaches in the Emergency Department. Cureus. 2022 Jan 19;14(1):e21428. doi: 10.7759/cureus.21428. eCollection 2022 Jan. PMID 35103222
- [Background] Rocha-Romero A, Roychoudhury P, Cordero RB, Mendoza ML. [Self-applied sphenopalatine ganglion block for postdural puncture headache: four case reports]. Braz J Anesthesiol. 2020 Sep-Oct;70(5):561-564. doi: 10.1016/j.bjan.2020.07.002. Epub 2020 Sep 16. PMID 33032805